CLINICAL TRIAL: NCT04574219
Title: Feasibility and Acceptability of Virtual Parental Presence on Induction of Anesthesia - Modernizing Solutions for Pediatric Anesthesia in Response to COVID-19
Brief Title: Virtual Parental Presence on Induction
Acronym: VPPIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0371
Record Dates: First submitted 2020-09-24; First posted 2020-10-05 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Anxiety; Surgery
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Feasibility/Acceptability (Other): This arm will be used to assess the feasibility and acceptability of using FaceTime during induction.
  Interventions: Other: Use of Facetime with child and parents during induction
- Coaching prior to surgery (Other)
  Interventions: Other: Use of Facetime with child and parents during induction
- Coaching day of surgery (Other)
  Interventions: Other: Use of Facetime with child and parents during induction

INTERVENTIONS:
Other: Use of Facetime with child and parents during induction — Families will be able to use Facetime with their child when the child is taken to the operating room

SUMMARY:
Our goal in this study is to investigate the feasibility and acceptability of virtual parental presence of parents on anxiety in children at induction of anesthesia at Cincinnati Children's Hospital, an institution whose use of parental presence on induction is deeply ingrained in our culture, and to determine the impact of coaching of parents either prior to arrival at the hospital vs. on the day of surgery on efficacy of virtual parental presence on induction. Our primary hypothesis is that virtual PPIA is both feasibile for the smooth induction of general anesthesia and is acceptable to parents, patients, and anesthesia providers at our isntutition. Our secondary hypothesis is that the coaching of parents prior to virtual PPIA enhances the effect of video parental presence at induction of anesthesia on children's anxiety and that coaching prior to arrival at the hospital will allow for increased ease and use of this technique.

ELIGIBILITY:
Inclusion Criteria:

* Children from ages 4 years to 12 years old
* ASA physical status I, II or III
* Planned inhalational induction
* Children presenting from home prior to surgery (not an inpatient)
* English speaking parents and child

Exclusion Criteria:

* children with developmental delay
* children with psychological / emotional disorders
* children with altered mental status
* children with language barrier
* children who are not accompanied by someone able to consent (ie legal guardian)
* children who are inpatient prior to surgery
* children with expected difficult intubation/airway
* children presenting for emergency surgery
* family history or personal history of malignant hyperthermia / risk of MH
* consent not obtained or withdrawl of consent
* children with past history of violent behaviors during induction of anesthesia
* cancellation of surgery
* patients with a diagnosis of COVID-19 or a patient under investigation for COVID-19, including patients being treated with airborne precuations in the operating room
* receipt of any type of medical sedative prior to induction of anesthesia, including (but not limited to) midazolam, ketamine, and/or dexmedetomidine.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Virtual presence cause delays in operating room | During procedure
  Based off operating room scheduled time vs actual start time
Parent satisfaction with virtual presence | Immediately after induction
  Parent will complete a satisfaction form which is 6 questions rating experience. Ratings are rated Excellent to Poor.
Operating room provider satisfaction | Immediately after procedure
  NASA Task Load Index questionnaire. The NASA task load index (NASA TLX) is a tool for measuring and conducting a subjective mental workload (MWL) assessment. It allows you to determine the MWL of a participant while they are performing a task. It rates performance across six dimensions to determine an overall workload rating.
Operating room provider satisfaction | Immediately after procedure
  System Usability Scale. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree.
Operating room induction nurse satisfaction | Immediately after procedure
  NASA Task Load Index questionnaire. The NASA task load index (NASA TLX) is a tool for measuring and conducting a subjective mental workload (MWL) assessment. It allows you to determine the MWL of a participant while they are performing a task. It rates performance across six dimensions to determine an overall workload rating.
Operating room induction nurse satisfaction | Immediately after procedure
  System Usability Scale. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree.
Assessment of parental presence with either Facetime, Skype or Teams | During patients induction, assessed immediately
  Parent and child will use one of three applications during the induction process

SECONDARY OUTCOMES:
Anxiety of child | Prior to induction
  Use of modified Yale Preoperative Anxiety Scale (mYPAS) measures anxiety at anesthesia induction. It looks at activity, facial expression, alertness and arousal, vocalization and interaction with adults.
Anxiety of child | During induction process, assessed immediately
  Use of modified Yale Preoperative Anxiety Scale (mYPAS) measures anxiety at anesthesia induction. It looks at activity, facial expression, alertness and arousal, vocalization and interaction with adults.
Child behavior induction compliance | During induction, assessed immediately
  Child Behavior Induction Assessment is an observational scale, used to describe the compliance of a child during induction of anesthesia.
Parent anxiety | Prior to patient moving to operating room
  State-Trait Anxiety Inventory assesses anxiety in adults. Responses are rated "Not at All" to "Very Much So"
Patient previous induction experience | After induction complete, assessed immediately
  Parent will complete form regarding previous experience. Will use a likert scale to compare previous experience to virtual presence experience
Parental Coaching - Prior | One week prior to surgery date
  Parents will review a standard video and handout for a week prior to surgery. Both will outline desired behaviors to support child during induction process.
Parental Coaching - Day | 1-2 hours before procedure
  Parents will review a standard video and handout the day of surgery. Both will outline desired behaviors to support child during induction process.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Goldschneider, MD, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (2):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States
- Hospital for Sick Children, Toronto, Ontario, Canada